CLINICAL TRIAL: NCT04720521
Title: Application of OpticalEnhancement Endoscopy（OE） in Diagnosis of Early Gastric Cancer: a Multicenter, Prospective, Randomized Controlled Study
Brief Title: Application of OE in Diagnosis of EGC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Collaborators: Qilu Hospital of Shandong University (Other); Shengjing Hospital (Other); Zhengzhou Central Hospital (Other); Shanghai Tongji Hospital, Tongji University School of Medicine (Other); Tang-Du Hospital (Other); Sino-Japanese Friendship Hospital of Jilin University (Unknown); First People's Hospital of Hangzhou (Other); Nanjing First Hospital, Nanjing Medical University (Other); Peking University Cancer Hospital & Institute (Other); The First People's Hospital of Guangzhou (Unknown); First Affiliated Hospital of Guangxi Medical University (Other); Tongji Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Director of Gastroenterology Dept, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: OE2021
Record Dates: First submitted 2021-01-20; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: High Risk Population of Gastric Cancer
Keywords: early gastric cancer; Optical Enhancement; Detection Rate
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OE+white light (Experimental): Using white light firstly to observe from esophagus to duodenum and then switch OE mode to observe from antrum to esophagus.
  Interventions: Diagnostic Test: OE+white light
- White light (No Intervention): Using White light to observe from esophagus to duodenum.

INTERVENTIONS:
Diagnostic Test: OE+white light — Firstly use white light to observe from esophagus to duodenum and then switch OE mode to observe from antrum to esophagus
  Arms: OE+white light

SUMMARY:
The main purpose of this study is to evaluate application value of OE mode 2 in the diagnosis of early gastric cancer The Secondary purpose is to evaluate application value of OE mode 1 in differentiating the diagnosis of neoplastic lesions of the gastric mucosa.

DETAILED DESCRIPTION:
Gastric cancer is the most prevalent cancer in China，while the detection rate of early gastric cancer is lower than 10%. An effective screening method to improve the detection rate is urgently needed. Optical Enhancement (OE) mode is an endoscopic mode that uses the principle of grating for electronic staining, which provides a clear picture of the submucosal and superficial mucosal vascular structures. The OE1 mode provides enhanced images of the gastric Gland tube and blood vessels, as well as magnification. The OE2 mode is used to identify small chromatic aberrations and to visualize superficial structures in the gastric mucosa. So we designed this randomized controlled trial to discuss effectiveness of OE in the diagnosis of early gastric cancer and we hope to find an effective method to improve the detection rate of early gastric cancer in China.

ELIGIBILITY:
Inclusion Criteria:

Meet item 1or 2 + any items of 3-7

1. Male ≥ 40 years old, female ≥ 50 years old.
2. More than one year since the last gastroscopy.
3. Patients from the areas with high incidence of stomach cancer (Shandong Province, Liaoning Province, Fujian Province, Gansu Province, Qinghai Province, Ningxia Province, Jilin Province, Jiangsu Province, Shanghai).
4. Patients with pre-cancerous gastric diseases such as chronic atrophic gastritis, gastric ulcer, gastric polyp, hypertrophic gastritis, pernicious anemia, etc. in the past.
5. First-degree relatives of patients with a family history of gastric cancer.
6. Other high-risk life factors for gastric cancer (high salt, pickled diet, smoking, heavy alcohol consumption, etc.)
7. Positive serum gastric function tests (GastroPanel) include: H. pylori (H.P) antibody （+）, Fasting pepsinogen I and II ratio (PG I/PGII) <3.89, gastrin 17 (G-17) >1.50 pmol/L.

Exclusion Criteria:

1. Patients who have undergone invasive treatment such as surgical resection, PEG, chemotherapy etc. of either stomach or oesophagus. (except for EMR and ESD).
2. Patients with a confirmed diagnosis of progressive cancer above T2 degreed according to the TMN classification of cancer。
3. Patients on anticoagulants that cannot be biopsied.
4. Patients who have undergone gastrectomy.
5. Patients who have taken PPIs or H2 receptor antagonist within two weeks.
6. Patients with history of malignant neoplasm; high suspicion of neoplasm; severe cardiac, pulmonary, hepatic or renal insufficiency; severe mental illness and pregnant women.
7. Patients who did not signed the consent form.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2454 (Estimated)
Dates: Start 2019-05-10 (Actual); Primary Completion 2021-03-10 (Estimated); Study Completion 2021-05-10 (Estimated)

PRIMARY OUTCOMES:
Detection rate of gastric neoplastic lesion | procedure
  Include early gastric cancer, high-grade neoplasia, low-grade neoplasia and adenoma

SECONDARY OUTCOMES:
Specificity of detecting gastric neoplastic lesion | procedure
Sensitivity of detecting gastric neoplastic lesion | procedure

CONTACTS AND LOCATIONS:
Overall Officials: Zhao shen Li, M.D., Principal Investigator — Department of Gastroenterology, Changhai Hospital, Second Military Medical University
Locations (1):
- Department of Gastroenterology, Changhai Hospital, Second Military Medical University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gomez JM, Wang AY. Gastric intestinal metaplasia and early gastric cancer in the west: a changing paradigm. Gastroenterol Hepatol (N Y). 2014 Jun;10(6):369-78. PMID 25013389
- [Result] Nagao M, Nishikawa J, Ogawa R, Sasaki S, Nakamura M, Nishimura J, Goto A, Hashimoto S, Okamoto T, Suenaga M, Hamamoto Y, Sakaida I. Evaluation of the Diagnostic Ability of Optical Enhancement System in Early Gastric Cancer Demarcation. Gastroenterol Res Pract. 2016;2016:2439621. doi: 10.1155/2016/2439621. Epub 2016 Sep 28. PMID 27774101